CLINICAL TRIAL: NCT06568003
Title: TRIal to Evaluate TraNsvenous TrIcuspid Valve ReplacemenT With LuX-Valve Plus System in Patients With Severe or Greater Tricuspid Regurgitation - SafetY and Clinical Performance
Brief Title: TraNsvenous TrIcuspid Valve ReplacemenT With LuX-Valve Plus System (TRINITY-US)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jenscare Innovation Inc. (Industry)
Collaborators: Cardiovascular Research Foundation, New York (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JSNL-CIP-TVS02-01FDA
Record Dates: First submitted 2024-08-15; First posted 2024-08-23 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Tricuspid Regurgitation (TR)
Keywords: Tricuspid Regurgitation; Transvenous Tricuspid Replacement; LuX-Valve Plus System
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- : LuX-Valve Plus transvenous tricuspid valve and delivery system(LuX-Valve Plus System) (Experimental): The LuX-Valve Plus System is intended for the treatment of patients with severe TR who are determined by a Heart Team to be at high risk of traditional open-heart surgery.
  Interventions: Device: Transcatheter Tricuspid Valve Intervention

INTERVENTIONS:
Device: Transcatheter Tricuspid Valve Intervention — Due to unsustainable effect of medical therapy and high risks of surgical treatment, transcatheter tricuspid valve intervention (TTVI) has been a major field of study in the world in the last 10 years. TTVI could potentially reduce TR with lower periprocedural risk and improve the patient's clinical status and prognosis. Per the ESC guidelines for surgical and interventional treatment of tricuspid regurgitation (2021 ESC/EACTS Guidelines for the Management of Valvular Heart Disease), Transcatheter intervention for symptomatic secondary severe TR may be considered in inoperable patients at a Heart Valve Centre with expertise in the treatment of tricuspid valve disease (Class IIb). 20 Transcatheter tricuspid treatment options can be divided into categories based on their mechanism of action: coaptation enhancement (edge-to-edge repair and spacer device), annuloplasty devices, caval valve implantation and valve replacement.

SUMMARY:
The LuX-Valve Plus System is intended for the treatment of patients with at least severe TR who are symptomatic and determined by a Heart Team not to be suitable for surgical treatment. This study aims to assess the safety and effectiveness of the LuX-Valve Plus System in high-surgical risk patients with at least severe tricuspid regurgitation (TR).

DETAILED DESCRIPTION:
Investigational Device:

The LuX-Valve Plus System consists of the following elements:

1. a bioprosthetic valve consistent of bovine pericardial tissue mounted on a self-expanding nitinol stent frame (hereafter referred to as LuX-Valve Implant).The LuX-Valve Implant consists of a trileaflet bovine-pericardial-tissue valve, a nitinol self-expanding stent, a fabric skirt, a pair of clips, an anchoring pin and sutures.
2. a catheter-based delivery system (hereafter referred to as LuX-Valve Delivery Device),
3. an Introducer Kit for transvenous access, and
4. a delivery system Stabilizer.

   * The LuX-Valve Implant sizes:

     o JS/TTVI-28-40, JS/TTVI-28-45, JS/TTVI-28-50, JS/TTVI- 28-55, JS/TTVI-30-40, JS/TTVI-30-45, JS/TTVI-30-50, JS/TTVI-30-55, JS/ TTVI-30-60, JS/TTVI-30-65
   * LuX--Valve Plus Delivery System

     o JS/TTVDJ-33
   * Introducer Kit

     o JS/SID01-33-100
   * Stabilizer o JS/STA-TJ01-01

Primary Objective:

To assess the safety and effectiveness of the LuX-Valve Plus System in patients with at least severe tricuspid regurgitation (TR) who are at high risk for surgical treatment.

Study Sites and Geography:

Up to 3 centers in the United States.

Number of Subjects:

Up to 15 subjects will be enrolled.

Indications for Use:

The LuX-Valve Plus System is intended for the improvement of health status in patients with at least severe TR who are symptomatic and determined by a Heart Team to be at high risk for surgical treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years at time of consent
* Severe or greater TR assessed on transthoracic echocardiography by Echocardiography Core Lab using a 5-grade classification (Mild, Moderate, Severe, Massive, Torrential).
* New York Heart Association (NYHA) Class II-IV
* The Patient is being treated on optimal dosage for diuretics at investigator discretion
* The Site Heart Team concur the patient is not an optimal candidate for surgical treatment and it is anatomically suitable for transcatheter tricuspid valve replacement
* Patient must be able to fully understand all aspects of the investigation that are relevant to the decision to participate and provide a written informed consent
* Anatomical inclusion criteria confirmed by echocardiographic core lab, CT core lab and Eligibility Committee

Exclusion Criteria:

* Left Ventricular Ejection Fraction (LVEF) <35%
* Pulmonary arterial systolic pressure (PASP) >60 mmHg by echo Doppler (unless right heart catheterization [RHC] demonstrates PASP ≤60mmHg); or Right heart catheterization OR PASP >2/3 systemic BP with PVR >5 Wood units after vasodilator challenge, in the absence of symptomatic hypotension or systolic BP <90 mmHg.
* Evidence of intracardiac mass, thrombus, or vegetation
* Ebstein Anomaly or congenital right ventricular dysplasia
* Surgical correction is indicated for other concomitant valvular disease (subjects with concomitant valvular disease may treat their respective valve first and wait 2 months before being reassessed for the trial)
* Patients with valve prostheses implanted in the tricuspid valve
* Pre-existing prosthetic valve(s) (other than tricuspid ones) with clinically significant prosthetic dysfunction
* Active infection, infective endocarditis or sepsis within 3 months, or infections requiring antibiotics treatment within two weeks prior to planned procedure
* Untreated clinically significant coronary artery disease requiring revascularization
* Acute myocardial infarction or unstable ischemia-related angina within 30 days prior to the planned procedure
* Any percutaneous coronary, intracardiac or carotid intervention within 30 days prior to the planned procedure
* Any coronary or intracardiac or carotid intervention within 30 days prior to the planned procedure
* Cardiogenic shock manifested by low cardiac output, vasopressor dependence, or mechanical hemodynamic support TRINITY-US Trial #: Ver 1.0, 14 Nov 2023, Confidential Page 7 of 8
* Cerebrovascular stroke (ischemic or bleeding) within prior 3 months to enrollment
* Active peptic ulcer or active gastrointestinal bleeding within prior 3 months to enrollment
* Blood dyscrasias as defined: leukopenia (WBC <1000 mm3), thrombocytopenia (platelet count <50,000 cells/mm3), history of bleeding diathesis, or coagulopathy
* Inability to tolerate anticoagulation or antiplatelet therapy
* Severe liver failure
* Renal insufficiency (eGFR <30 mL/min [per the Cockcroft-Gault formula] and/or renal replacement therapy)
* Uncontrolled atrial fibrillation (e.g., resting heart rate >120 bpm)
* Pregnancy or intent to become pregnant prior to completion of all protocol follow-up requirements
* Severe Chronic Obstructive Pulmonary Disease requiring steroids or requiring continuous home oxygen
* Untreatable hypersensitivity or contraindication to any of the following: all antiplatelets, all anticoagulants, nitinol alloys (nickel and titanium), bovine tissue, glutaraldehyde, or contrast media
* Estimated life expectancy <12 months.
* Subjects currently participating in another clinical trial of an investigational drug or device that has not yet completed its primary endpoint
* Patients with current history of illicit drug use
* Any other condition making it unlikely the patient will be able to complete all protocol procedure and follow-ups determined by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-09-26 (Actual); Primary Completion 2025-10-02 (Actual); Study Completion 2030-10 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome - Post-procedural TR Remission Rate | at 30 days post procedure
  Defined as: Post-procedural TR of moderate or less (TR≤2+) without clinically significant paravalvular leak (PVL) on a transthoracic echocardiography (TTE) at 30 days post- procedure (Assessed by the Echocardiography Core Lab using a 5-grade classification)
Primary Outcome - Incidence of major adverse events at 30 days post procedure | at 30 days post procedure
  A composite endpoint of Major Adverse Event (MAE) at 30 days post procedure, as listed below:
  * Cardiovascular Death
  * Myocardial Infarction (MI)
  * Stroke
  * New Onset Renal Failure Requiring Unplanned Dialysis or Hemofiltration
  * Major Bleeding (includes type 3b or higher as defined by Tricuspid Valve Academic Research Consortium [TVARC])
  * Tricuspid Valve Surgery or Transcatheter Re-intervention post Procedure
  * Major Access Site and Vascular Complications
  * Major Cardiac Complications
  * Device-related Pulmonary Embolism
  * New Pacemaker Implantation due to Atrioventricular (AV) Block

SECONDARY OUTCOMES:
Acute Secondary Endpoints - Intraprocedural success Rate | the first 24h post-procedure
  Subjects in whom all of the following were present were considered intraprocedural success, otherwise they were considered intraprocedural failure:
  * Absence of intraprocedural mortality or stroke; and
  * Successful access, delivery, and retrieval of the device delivery system
  * Successful deployment and correct positioning of the intended device without requiring implantation of unplanned additional device
  * Adequate performance of the transcatheter device. Absence of tricuspid stenosis (TVA ≥1.5cm2 or TVAi≥0.9cm2/m2), DVI<2.2, mean gradient <5mmHg; reduction of total tricuspid regurgitation to acceptable (moderate [2+])
  * Absence of device-related obstruction of forward flow
  * Absence of device-related pulmonary embolism
  * Freedom from emergency surgery or reintervention during the first 24h related to the device or access procedure
Acute Secondary Endpoints - Clinical success Rate | at 30 days and at 1 year post-procedure
  Subjects in whom all of the following were present were considered clinical success:
  * Absence of procedural mortality and stroke
  * Proper position of the device with adequate performance of the transcatheter device. Absence of tricuspid stenosis (TVA≥1.5cm2 or TVAi≥0.9cm2/m2), DVI<2.2, mean gradient<5mmHg; reduction of total tricuspid regurgitation to moderate [2+]
  * Freedom from unplanned surgical or interventional procedures related to the device or access procedure
  * Absence of MAEs, including:
    1. Life-threatening bleeding (TVARC 5)
    2. Major vascular complications
    3. Major cardiac structural complications
    4. Stage 2 or 3 acute kidney injury (includes new dialysis)
    5. Myocardial infarction or coronary ischemia requiring percutaneous coronary intervention or coronary artery bypass graft.
    6. Device-related obstruction of forward flow
    7. Device-related pulmonary embolism
    8. Hemodynamic compromise leading to heart transplantation or major cardiac

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Henry Ford Health System, Detroit, Michigan
  - Montefiore Medical Center, New York, New York